CLINICAL TRIAL: NCT01231776
Title: Study of Acupuncture of Traditional Chinese Medicine
Brief Title: Acupuncture Improves Sleep in Patients Undergoing Cardiopulmonary Bypass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: zhang jinzhou, the departement of cardiovascular surgery, xijing hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20100926
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2010-09

CONDITIONS: Heart Valve Diseases; Cardiopulmonary Bypass
Keywords: cardiopulmonary bypass; sleep; acupuncture
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control group (No Intervention)
  Interventions: Other: electronic acupuncture
- acupuncture preoperative (Active Comparator): acupuncture before operation for one week
  Interventions: Other: electronic acupuncture
- acupuncture in hospital (Active Comparator): acupuncture all the time in hospital
  Interventions: Other: electronic acupuncture

INTERVENTIONS:
Other: electronic acupuncture — applying a stimula on neiguang and shenmen through electronic acupuncture

SUMMARY:
Due to various causes, such as brain impairment, environment changes, anxious,et al. patients, who undergo cardiopulmonary bypass, often suffer from poor quality of sleep. In chinese traditional medicine, acupuncture can improve the quality of sleep in patients with sleeping disorder. But it remains acupuncture could improve the quality of sleep in patients with heart operations.

DETAILED DESCRIPTION:
60 patients are divided into three groups. control group: no any intervention; experiment group 1: acupuncture are used in patients before cardiac operation; experiment group 2: acupuncture are used through all the course in hospital.

before operation, before discharge, one month after operation, two month after operation, the quality of sleep are evaluated. and comparisons will be made in three groups.

ELIGIBILITY:
Inclusion Criteria:

* aging:18yr--65yr
* cardiopulmonary bypass
* NYHA ≤II and EF≥50%
* not illiterate person

Exclusion Criteria:

* neurological disease,mentality disorder
* abuse of alcohol
* long history of smoking
* sleep disorder before admitting to hospital

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-01 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
multiple monitoring for sleeping | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: zhang jinzhou, MD, Principal Investigator — Xijing Hospital
Locations (1):
- Zhang Jinzhou, Xi'an, Shaanxi, China